CLINICAL TRIAL: NCT01188993
Title: Hemodynamic Assessment With Transpulmonary Thermodilution and Transesophageal Echocardiography in Patients With Early Septic Shock
Brief Title: Transpulmonary Thermodilution and Transesophageal Echocardiography in Early Septic Shock
Acronym: HEMOSEPSIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I09003
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2010-08

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- septic shock TPT then TEE (Active Comparator): Group 1: Each patient will be assessed by both the transpulmonary thermodilution technique and transesophageal echocardiography (TEE)..
  Interventions: Combination Product: early septic shock
- septic shock TEE then TPT (Active Comparator): Goup 2: Each patient will be assessed by both transesophageal echocardiography (TEE) and the transpulmonary thermodilution technique.
  Interventions: Combination Product: early septic shock

INTERVENTIONS:
Combination Product: early septic shock — Each patient will be assessed by both the transpulmonary thermodilution and Transesophageal Echocardiography.

SUMMARY:
The purpose of this study is to assess the concordance of therapeutic changes proposed after an early hemodynamic evaluation (hemodynamic profile) in septic shock patients using jointly the transpulmonary thermodilution technique and transesophageal echocardiography (TEE).

DETAILED DESCRIPTION:
Each patient will be assessed by both the transpulmonary thermodilution technique and TEE (H0). The two assessments will be performed in random order (central randomization stratified by participating center), but within 30 minutes (no change of ongoing treatment during the assessment period). Two investigators not involved in patient care and blinded to the results of the alternative technique will performed independently the hemodynamic assessment using one of the two modalities for hemodynamic assessment tested in the study. They will interpret the results at bedside and propose a therapeutic change to the attending physician, according to the hemodynamic profile. The latter will finally: precisely identify the clinical problem to be solved (e.g., therapeutic target of the Surviving Sepsis Campaign not reached, tissue hypoperfusion), choose a therapy adapted while taking into account the clinical scenario and the results of both the transpulmonary thermodilution and TEE, evaluate the efficacy of this treatment (problem solved or not) and its tolerance (potential side-effect attributable to the treatment). In addition, the presence or resolution of signs of tissue hypoperfusion will systematically be assessed at H6, H12 and H24. Primary and secondary outcomes will be assessed by an independent committee of experts.

ELIGIBILITY:
Inclusion Criteria:

* ventilated patient in sinus rhythm with septic shock requiring a hemodynamic assessment

Exclusion Criteria:

* < 18 yr-old
* pregnancy
* contra-indication for TEE, non sinus rhythm, aplasia, prior participation to the study, hemodynamic assessment using any other technique than those tested in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
therapeutic procedure following the hemodynamic assessment | 2 years
  Changes in therapy proposed after the hemodynamic assessment (hemodynamic profile) by each of the two tested methods: blood volume expansion (preload responsiveness), positive inotrope (cardiac dysfunction), vasopressor (vasoplegia), no change in ongoing therapy or dose tapering (inotropes or vasopressor).

SECONDARY OUTCOMES:
efficacy and safety of therapeutic intervention | 2 years
  Efficacy (clinical problem solved) and tolerance (potential side-effects) of the therapeutic change.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Bordeaux UH, Bordeaux
  - Toulouse UH, Toulouse

REFERENCES:
- [Result] Vignon P, Begot E, Mari A, Silva S, Chimot L, Delour P, Vargas F, Filloux B, Vandroux D, Jabot J, Francois B, Pichon N, Clavel M, Levy B, Slama M, Riu-Poulenc B. Hemodynamic Assessment of Patients With Septic Shock Using Transpulmonary Thermodilution and Critical Care Echocardiography: A Comparative Study. Chest. 2018 Jan;153(1):55-64. doi: 10.1016/j.chest.2017.08.022. Epub 2017 Sep 1. PMID 28866112